CLINICAL TRIAL: NCT04555720
Title: The Benchmark Clinic: An Interdisciplinary Comprehensive Care Model for People With Parkinson Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00105281
Record Dates: First submitted 2020-09-14; First posted 2020-09-21 (Actual); Results first posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2022-04

CONDITIONS: Parkinson Disease
Keywords: interdisciplinary care; patient engagement; preventative care
MeSH Terms: conditions — Parkinson Disease; Patient Participation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interdisciplinary Care (Experimental): If assigned to the interdisciplinary group, participants will see social work, physical therapy, occupational therapy, speech therapy, and pharmacy in a scheduled rotation for about 45 minutes each. After these evaluations, the team meets with the participant's doctor for a discussion of treatment. After this meeting, the participants doctor will meet to discuss a treatment plan and make recommendations.
  Interventions: Behavioral: Interdisciplinary Visit
- Standard of Care (No Intervention): If assigned to standard of care, group participants will have a normally scheduled visit with neurologist.

INTERVENTIONS:
Behavioral: Interdisciplinary Visit — If assigned to the interdisciplinary group, participants will see social work, physical therapy, occupational therapy, speech therapy, and pharmacy in a scheduled rotation for about 45 minutes each. After these evaluations, the team meets with the participants doctor for a discussion of treatment. After this meeting, the participants doctor will meet to discuss a treatment plan and make recommendations.
  Arms: Interdisciplinary Care

SUMMARY:
The purpose of this study is to determine if an interdisciplinary clinic can help people with Parkinson's disease care for themselves, improve their ability to follow recommended treatments, and have fewer problems like falls or visits to the emergency room.

Participants will be randomly assigned to receive either care from the interdisciplinary clinic or standard neurological specialist care.

This study involves questionnaires both before and 3 months after participation in a one time interdisciplinary care clinic or standard care depending on which type of care the participant is randomized to. Participants will be in the study for up to 6 months. The study will end upon completion of questionnaires about 3 months after treatment with the interdisciplinary care clinic or standard care.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Parkinson's Disease over the age of 30,
* Caregiver willing to also participate.
* Must be able to provide consent.

Exclusion Criteria:

-Atypical Parkinsonism

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2021-02-03 (Actual); Primary Completion 2021-09-28 (Actual); Study Completion 2021-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyle Mitchell, MD, Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Interdisciplinary Care - Caregivers: Caregivers for participants in the Interdisciplinary Care arm
- Standard of Care - Caregivers: Caregivers for participants in the standard of care arm
Period: Overall Study
Arm/Group | Interdisciplinary Care | Standard of Care | Interdisciplinary Care - Caregivers | Standard of Care - Caregivers
Started | 24 | 25 | 7 | 5
Completed | 18 | 19 | 7 | 5
Not Completed | 6 | 6 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 6 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Only participants in the Interdisciplinary Care and Standard of Care Arms who completed the study are included. Baseline demographic information was not collected from the 2 Caregiver Arms.
Groups:
- Total: Total of all reporting groups
Arm/Group | Interdisciplinary Care | Standard of Care | Interdisciplinary Care - Caregivers | Standard of Care - Caregivers | Total
Number analyzed (Participants) | 18 | 19 | 0 | 0 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age of participants in the 2 Caregiver arms was not collected
  years | 66.9 (10.2) | 62.5 (10.4) |  |  | 64.6 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Sex was not collected for participants in the 2 Caregiver arms
  Participants
    Female | 6 | 7 | 0 | 0 | 13
    Male | 12 | 12 | 0 | 0 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Ethnicity of participants in the 2 Caregiver arms was not collected
  Participants
    Hispanic or Latino | 0 | 1 |  |  | 1
    Not Hispanic or Latino | 18 | 18 |  |  | 36
    Unknown or Not Reported | 0 | 0 |  |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Race of participants in the 2 Caregiver Arms was not collected
  Participants
    American Indian or Alaska Native | 0 | 0 |  |  | 0
    Asian | 0 | 1 |  |  | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 |  |  | 0
    Black or African American | 0 | 3 |  |  | 3
    White | 18 | 15 |  |  | 33
    More than one race | 0 | 0 |  |  | 0
    Unknown or Not Reported | 0 | 0 |  |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 18 | 19 |  |  | 37

OUTCOME MEASURES:

1. Primary Outcome: Change in Composite Score on Self-efficacy Scale
Description: Title of scale: Self-efficacy Scale for Chronic Diseases. This is a validated scale. Minimum score is 6, Maximum score is 60. Higher score is a better outcome.
Time Frame: Baseline, 3 months after interdisciplinary or standard clinic visit
Population: Data was not collected for the "Interdisciplinary Care - Caregivers" and "Standard of Care - Caregivers" groups.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Interdisciplinary Care | Standard of Care
Number analyzed (Participants) | 18 | 19
score on a scale | 38.5 [30 to 42] | 43 [38 to 49]

2. Secondary Outcome: Change in Total Weekly Minutes Exercised as Measured by Patient Engagement Survey.
Description: Investigator developed patient engagement survey
Time Frame: Baseline, 3 months after interdisciplinary or standard care visit
Population: Data was not collected for the "Interdisciplinary Care - Caregivers" and "Standard of Care - Caregivers" groups.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Interdisciplinary Care | Standard of Care
Number analyzed (Participants) | 18 | 19
minutes | 138.3 (186.4) | 205.2 (147)

3. Secondary Outcome: Change in Caregiver Burden Score on Zarit Burden Interview Scale
Description: Title of scale: Zarit Burden Interview. This is validated scale. Minimum score is 0. Maximum score is 88. Higher score is a worse outcome.
Time Frame: Baseline, 3 months after interdisciplinary or standard care visit
Population: Only care partners were analyzed
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Interdisciplinary Care - Caregivers | Standard of Care - Caregivers
Number analyzed (Participants) | 7 | 5
score on a scale | 8 [5 to 16] | 16 [9 to 17]

4. Secondary Outcome: Number of Skilled Therapy Visits as Reported by Participant
Description: Number of skilled therapy visits as reported by participant
Time Frame: Baseline, 3 months after interdisciplinary or standard care visit
Population: Data was not collected for the "Interdisciplinary Care - Caregivers" and "Standard of Care - Caregivers" groups.
Measure: Mean (Standard Deviation); unit: visits
Arm/Group | Interdisciplinary Care | Standard of Care
Number analyzed (Participants) | 18 | 19
visits | 3.5 (8.5) | 9 (23.1)

5. Secondary Outcome: Number of Participants With a Hospitalization as Reported by Participant and Medical Record Review
Description: Number of participants with a hospitalization as reported by participant and medical record review
Time Frame: Baseline, 3-6 months after interdisciplinary or standard care visit
Population: Data was not collected for the "Interdisciplinary Care - Caregivers" and "Standard of Care - Caregivers" groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Interdisciplinary Care | Standard of Care
Number analyzed (Participants) | 18 | 19
Participants | 1 | 8

6. Secondary Outcome: Number of Participants With an ER Visit as Reported by Participant and Medical Record Review
Description: Number of participants with an ER visit as reported by participant and medical record review
Time Frame: Baseline, 3-6 months after interdisciplinary or standard care visit
Population: Data was not collected for the "Interdisciplinary Care - Caregivers" and "Standard of Care - Caregivers" groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Interdisciplinary Care | Standard of Care
Number analyzed (Participants) | 18 | 19
Participants | 5 | 11

7. Secondary Outcome: Number Participants With a Fall as Reported by Participant and Medical Record Review
Description: Number participants with a fall as reported by Participant and Medical Record Review
Time Frame: Baseline, 3 months after interdisciplinary or standard care visit
Population: Data was not collected for the "Interdisciplinary Care - Caregivers" and "Standard of Care - Caregivers" groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Interdisciplinary Care | Standard of Care
Number analyzed (Participants) | 18 | 19
Participants | 3 | 2

8. Secondary Outcome: Number of Participants With a Contraindicated Medication Combination as Determined by Medical Record Review
Description: Number of participants with a contraindicated medication combination as determined by medical record review
Time Frame: Baseline, 3-6 months after interdisciplinary or standard care visit
Population: Data was not collected for the "Interdisciplinary Care - Caregivers" and "Standard of Care - Caregivers" groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Interdisciplinary Care | Standard of Care
Number analyzed (Participants) | 18 | 19
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Within 3 months of clinic visit
Description: Self-report. Adverse events were not collected for the 2 Caregiver Arms.
Arm/Group | Interdisciplinary Care | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/19
Other Adverse Events (participants affected / at risk) | 0/18 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-01-29): https://cdn.clinicaltrials.gov/large-docs/20/NCT04555720/Prot_SAP_000.pdf
  • Informed Consent Form (2020-09-16): https://cdn.clinicaltrials.gov/large-docs/20/NCT04555720/ICF_001.pdf